CLINICAL TRIAL: NCT02473445
Title: A Long-Term Open-Label Extension Study of RP103-MITO-001 to Assess the Safety, Tolerability and Efficacy of Cysteamine Bitartrate Delayed-release Capsules (RP103) for Treatment of Children With Inherited Mitochondrial Disease
Brief Title: A Long-term Extension of Study RP103-MITO-001 (NCT02023866) to Assess Cysteamine Bitartrate Delayed-release Capsules (RP103) in Children With Inherited Mitochondrial Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to end development of RP103 for mitochondrial disease due to lack of efficacy demonstrated in base study RP103-MITO-001.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP103-MITO-002
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Mitochondrial Diseases
Keywords: Inherited mitochondrial disease; Leigh Syndrome; Leber's Hereditary Optic Neuropathy (LHON); Myoclonic epilepsy and ragged-red fibers (MERFF); Mitochondrial encephalomyopathy, lactic acidosis, and stroke-like syndrome (MELAS); Kearn-Sayre syndrome; Polymerase gamma (POLG) -related disorders; Mitochondrial neurogastrointestinal encephalopathy syndrome (MNGIE)
MeSH Terms: conditions — Mitochondrial Diseases; Leigh Disease; Optic Atrophy, Hereditary, Leber; Epilepsies, Myoclonic; Mitochondrial Encephalomyopathies; Acidosis, Lactic; Ophthalmoplegia, Chronic Progressive External; Visceral myopathy familial external ophthalmoplegia | interventions — Cysteamine

STUDY DESIGN:
Intervention Model Description: Open-label extension study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysteamine Bitartrate Delayed-release (Experimental): Participants received cysteamine bitartrate delayed-release capsules (RP103) twice daily for up to 2 years. The starting dose was the same as the last dose received in study RP103-MITO-001, the maximum dose was 1.3 g/m²/day.
  Interventions: Drug: Cysteamine Bitartrate

INTERVENTIONS:
Drug: Cysteamine Bitartrate — Cysteamine Bitartrate Delayed-release capsules
  Other Names: RP103; PROCYSBI®

SUMMARY:
A long-term extension study to assess the safety, tolerability and efficacy of cysteamine bitartrate delayed-release capsules (RP103) in children with inherited mitochondrial diseases who previously enrolled into study RP103-MITO-001 (NCT02023866).

DETAILED DESCRIPTION:
Patients with inherited mitochondrial diseases associated with nuclear or mitochondrial deoxyribonucleic acid (DNA) mutations that impair the respiratory chain. These include, but are not limited to the following clinical syndromes: Leber's hereditary optic neuropathy; myoclonic epilepsy and ragged-red fibers (MERFF); mitochondrial encephalomyopathy, lactic acidosis, and stroke-like syndrome (MELAS); Kearn-Sayre syndrome; subacute necrotizing encephalopathy (Leigh Syndrome); polymerase gamma (POLG)-related disorders (Alpers-Huttenlocher Syndrome, Autosomal Dominant Progressive External Ophthalmoplegia, Autosomal Recessive Progressive External Ophthalmoplegia, Childhood Myocerebrohepatopathy Spectrum Disorders, Myoclonic Epilepsy Myopathy Sensory Ataxia, POLG-Related Ataxia Neuropathy Spectrum Disorders); Mitochondrial neurogastrointestinal encephalopathy syndrome (MNGIE), also called myoneurogastrointestinal encephalopathy syndrome or polyneuropathy-ophthalmoplegia-leukoencephalopathy- Intestinal pseudoobstruction (POLIP) syndrome; others, e.g., mitochondrial cardiomyopathies and other syndromes due to multiple mitochondrial DNA deletions.

Patients completing study RP103-MITO-001 (NCT02023866) are eligible for enrollment into the extension study RP103-MITO-002 if all inclusion and exclusion criteria are fulfilled. Subjects continue on the last total daily dose of cysteamine bitartrate delayed-release capsules taken during RP103-MITO-001. Dose-adjustments are permitted.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Completed all visits in Study RP103-MITO-001 (NCT02023866).
2. Body weight ≥ 5 kg.
3. The subject must be willing to abstain from initiating dietary supplements and non-prescribed medications except as allowed by the Investigator, throughout the study (from Day 1 to Study Exit).
4. Willing and able to comply with study drug dosing requirements, i.e. ingest the RP103 capsules intact, or sprinkled in liquid or soft food, or using a G-tube.
5. Sexually active female subjects of childbearing potential (i.e., not surgically sterile [tubal ligation, hysterectomy, or bilateral oophorectomy]) must agree to utilize two of the following acceptable forms of contraception throughout the study (from Day 1 to Study Exit):

   * Hormonal contraception: birth control pills, injection, patch, vaginal ring or implant;
   * Condom or diaphragm, with spermicide;
   * Intrauterine device (IUD);
   * Sterile male partner (vasectomy performed at least 6 months prior to the study).
6. Patient's legally authorized representative must provide written informed consent; Patient must provide assent, if required by local/institutional requirements.

Exclusion Criteria:

1. Documented diagnosis of concurrent inborn errors of metabolism.
2. Platelet count, lymphocyte count or hemoglobin below the lower limit of normal (LLN) at the Baseline visit.
3. Hepatic insufficiency with liver enzyme tests (alkaline phosphatase, aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than 2.5 times the upper limit of normal (ULN) at the Baseline Visit.
4. Bilirubin > 1.2 g/dL at the Baseline Visit.
5. Inability to complete the elements of the study, e.g., coma, hemodynamic instability or requiring continuous ventilator support.
6. Malabsorption requiring total parenteral nutrition (TPN), chronic diarrhea, bouts of pseudo obstruction.
7. Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis.
8. Patients with suspected elevated intracranial pressure, pseudotumor cerebri (PTC) and/or papilledema.
9. Severe gastrointestinal disease including gastroparesis.
10. History of drug or alcohol abuse.
11. History of pancreatitis.
12. Participated in an investigational drug trial (except the RP103-MITO-001 study) within 30 days or, within 90 days for a biologic, device, or surgical treatment, for inherited mitochondrial diseases prior to the Baseline Visit.
13. Known or suspected hypersensitivity to cysteamine and penicillamine.
14. Female subjects who are nursing, planning a pregnancy, known or suspected to be pregnant, or with a positive serum pregnancy test at the Baseline visit.
15. Patients who, in the opinion of the Investigator, are not able or willing to comply with the protocol.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - University of California at San Diego (UCSD), San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Akron Children's Hospital, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bousquet M, Gibrat C, Ouellet M, Rouillard C, Calon F, Cicchetti F. Cystamine metabolism and brain transport properties: clinical implications for neurodegenerative diseases. J Neurochem. 2010 Sep;114(6):1651-8. doi: 10.1111/j.1471-4159.2010.06874.x. Epub 2010 Aug 19. PMID 20569301
- [Background] Salmi H, Leonard JV, Rahman S, Lapatto R. Plasma thiol status is altered in children with mitochondrial diseases. Scand J Clin Lab Invest. 2012 Apr;72(2):152-7. doi: 10.3109/00365513.2011.646299. Epub 2012 Jan 2. PMID 22208644
- [Background] Maher P, Lewerenz J, Lozano C, Torres JL. A novel approach to enhancing cellular glutathione levels. J Neurochem. 2008 Nov;107(3):690-700. doi: 10.1111/j.1471-4159.2008.05620.x. Epub 2008 Aug 12. PMID 18702664
- [Background] Mancuso M, Orsucci D, Logerfo A, Rocchi A, Petrozzi L, Nesti C, Galetta F, Santoro G, Murri L, Siciliano G. Oxidative stress biomarkers in mitochondrial myopathies, basally and after cysteine donor supplementation. J Neurol. 2010 May;257(5):774-81. doi: 10.1007/s00415-009-5409-7. Epub 2009 Dec 4. PMID 19960200

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed study RP103-MITO-001 (NCT02023866) study were eligible for enrollment into this extension study. The study was conducted at 5 sites in the United States.
Period: Overall Study
Arm/Group | Cysteamine Bitartrate Delayed-release
Started | 22
Completed | 0
Not Completed | 22
Not completed — Withdrawal by Subject | 2
Not completed — Sponsor Decision | 20

BASELINE CHARACTERISTICS:
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Black of African American | 0
  Native Hawaiian or other Pacific Islander | 0
  White | 18
  Other | 0
  Multiple | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) Score
Description: The NPMDS evaluates the progression of mitochondrial disease in pediatric patients in 4 domains:
  I - Current Function (vision, hearing, communication, feeding, and mobility) with scores ranging from 0 to 21;
  II - System Specific Involvement (seizures, encephalopathy, bleeding diathesis or coagulation defects, gastrointestinal, endocrine, respiratory, cardiovascular, renal, liver, and blood) with scores ranging from 0 to 30.
  III - Current Clinical Assessment (growth and development over past 6 months, vision, strabismus and eye movement, myopathy, ataxia, pyramidal, extrapyramidal, and neuropathy) with scores ranging from 0 to 28;
  IV - Quality of Life with scores ranging from 0 to 25. For sections I-III, higher scores reflect more severe disease. For Section IV, a higher score reflects a lower quality of life.
Time Frame: Baseline, every 3 months and Study Exit (up to 24 Months)
Population: The study was closed prematurely due to lack of efficacy demonstrated in base study RP103-MITO-001. As a result, only a limited amount of data was collected for patients that were enrolled prior to termination. The decision was made that the data were not complete enough, and no analyses were conducted.
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 0

2. Secondary Outcome: Change Over Time in Two of the Most Pre-eminent Symptoms
Description: The two pre-eminent symptoms previously identified in study RP103-MITO-001 were to be continued to be assessed during the extension study. Symptoms included myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision.
Time Frame: Baseline, every 3 months and Study Exit (up to 24 Months)
Population: as for outcome 1
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 0

3. Secondary Outcome: Change Over Time in Pharmacodynamic Biomarkers
Description: Change from baseline in glutathione, glutathione disulfide, and lactate analyses were not performed as the study was prematurely terminated.
Time Frame: Baseline, every 3 months and Study Exit (up to 24 Months)
Population: as for outcome 1
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until the last dose; median duration of treatment was 238 days.
Arm/Group | Cysteamine Bitartrate Delayed-release
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 9/22
Other Adverse Events (participants affected / at risk) | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cysteamine Bitartrate Delayed-release (N=22)
Blepharospasm (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Clostridium difficile infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Muscle spasticity (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cysteamine Bitartrate Delayed-release (N=22)
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 5
Ataxia (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Myoclonus (Nervous system disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
The study was closed prematurely due to lack of efficacy demonstrated in base study RP103-MITO-001 and no efficacy analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .

DOCUMENTS (2):
  • Study Protocol (2014-12-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT02473445/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT02473445/SAP_001.pdf